CLINICAL TRIAL: NCT05447910
Title: Comprehensive Single-Cell Transcriptional Analysis of Aromatase Inhibitor-Resistant Breast Cancer
Brief Title: Analysis of Letrozole in Patients With Operable Hormone Receptor Positive, HER2 Negative Breast Cancer
Status: Terminated | Type: Observational
Why Stopped: insufficient funding
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 21-003046; NCI-2022-04802 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2022-06-28; First posted 2022-07-07 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Breast Adenocarcinoma; Invasive Breast Carcinoma; Resectable Breast Carcinoma
MeSH Terms: interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples store for future research with consent of participants
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with early-stage hormone receptor-positive HER2-negative breast cancer receiving letrozole: Patients undergo collection of blood and tissue samples prior to beginning treatment with letrozole and at least two weeks after the start of letrozole treatment, but prior to surgery.
  Interventions: Procedure: Biospecimen Collection

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood and tissue samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection

SUMMARY:
The purpose of this study is to study to collect tissue samples from patients with early stage hormone receptor-positive HER2-negative breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal and suitable to receive aromatase inhibitor as per physician's discretion
* Histologically confirmed un-resected operable invasive adenocarcinoma of the breast ≥ 0.5 cm with estrogen receptor (ER) and/or progesterone receptor (PR) positive ≥ 10%, and no human epidermal growth factor receptor 2 (HER2) amplification or overexpression
* Patients must not have received any prior chemotherapy, radiation therapy, or endocrine therapy for their current breast cancer. Patients who received tamoxifen or raloxifene or another agent for prevention of breast cancer may be included
* Willing and able to provide research tissue samples
* Willing and able to provide research blood samples

Exclusion Criteria:

* Immunocompromised patients including patients known to be human immunodeficiency virus (HIV) positive or those on chronic steroids

  * NOTE: Must be off systemic steroids at least 14 days prior to pre-registration. However, topical steroids, inhalants or steroid eye drops are permitted
* Known history of active autoimmune disease that has required systemic treatment within =< 30 days (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs) prior to pre-registration

  * NOTE: Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment. Patients with vitiligo, Graves disease, or psoriasis not requiring systemic treatment within the past 30 days are not excluded. Patients with Celiac disease controlled with diet modification are not excluded

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with early-stage hormone receptor-positive HER2-negative breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2022-07-21 (Actual); Primary Completion 2023-09-27 (Actual); Study Completion 2023-09-27 (Actual)

PRIMARY OUTCOMES:
Differences in tumor microenvironment subpopulations in aromatase inhibitor (AI)-sensitive version (vs.) AI-resistant hormone receptor (HR)+ breast cancer | Up to 8 weeks
  Tissue samples from patients with early-stage hormone receptor-positive HER2-negative breast cancer will be collected to compare differences.

SECONDARY OUTCOMES:
Effects of estrogen deprivation on the immune microenvironment | Up to 8 weeks
  Estrogen receptor will be evaluated by both biopsy and surgical specimens.
Effects of estrogen deprivation on tumor immune microenvironment | Up to 8 weeks
  Estrogen receptor will be evaluated by both biopsy and surgical specimens.

CONTACTS AND LOCATIONS:
Overall Officials: Saranya Chumsri, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-12-01): https://cdn.clinicaltrials.gov/large-docs/10/NCT05447910/Prot_SAP_000.pdf
  • Informed Consent Form (2023-05-08): https://cdn.clinicaltrials.gov/large-docs/10/NCT05447910/ICF_001.pdf